CLINICAL TRIAL: NCT01343641
Title: A Phase 2, Investigator-Initiated, Randomized, Double-Blind, Placebo-Controlled Study to Determine Growth Hormone Secretagogue MK-0677's Effect on Lean Body Mass in Chronic Kidney Disease Subjects With Stage 4 and Stage 5 Kidney Disease
Brief Title: Growth Hormone Secretagogue MK-0677's Effect on Lean Body Mass in Chronic Kidney Disease Stage 4/5 Subjects
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Could not obtain drug supply from manufacturer
Sponsor: University of Virginia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Warren K Bolton, MD, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 13684; NIH Grant Number-R21DK077372; IND Number-54,041
Record Dates: First submitted 2010-07-29; First posted 2011-04-28 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2012-04

CONDITIONS: Chronic Kidney Disease; Kidney Disease
Keywords: Kidney Disease; Chronic Kidney Disease; Growth Hormone
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases | interventions — ibutamoren mesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MK-0677 (Experimental): The oral agent MK-677 is spiropiperidine, Merck L-163 191, GH secretagogue ghrelin mimetic which increases GH and IGF-I secretion, fat free mass and energy expenditure76-79. It is produced by Merck & Co, Inc.
  Interventions: Drug: MK-0677
- Placebo (Placebo Comparator): Inactive Pill used as a comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK-0677 — The oral agent MK-677 is spiropiperidine, Merck L-163 191, GH secretagogue ghrelin mimetic which increases GH and IGF-I secretion, fat free mass and energy expenditure76-79. It is produced by Merck & Co, Inc.
  Arms: MK-0677
Drug: Placebo — Inactive Pill used as a comparator
  Arms: Placebo

SUMMARY:
This year-long investigator-initiated study is designed to determine effects of MK-0677, a GH secretagogue, in renal patients. It is a double-blind, placebo-controlled trial employing the following procedures: Informed consent process, followed by evaluation and screening tests to confirm patients' eligibility. Patients whose screening laboratory results for glycated hemoglobin level, thyroid function, or liver function exceed protocol eligibility criteria will not be randomized. Other exclusions are Congestive Heart Failure Class III or IV by the New York Heart Assocation's (NYHA) Guidelines and specified cardiovascular disorders within six months of baseline visit and muscle weakness associated with neuromuscular or neurological disorders. Before the subject begins taking the experimental drug MK-0677 or placebo, baseline assessments of subjects' hormone and cytokine levels, physical condition, body mass (determined by a DEXA scan), strength and functionality, and appetite will be obtained. In addition, quality of life assessments (SF-36) will be administered. This study's primary outcome is an increase in lean body weight. Secondary outcomes are cytokine and hormone levels, including, leptin, insulin, ghrelin, TNF- alpha, CRPs, IL-1, IL-6, and IL-10, ghrelin associated esterase and adiponectin, nutritional status, quality of life (QoL), food appreciation, physical function and economic impact. 70 subjects will be the enrollment target. This number was determined to offset projected screen failure and early withdrawal rates, and to ensure that 42 subjects complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18 to 85.
* GFR by the MDRD estimate ≤ 30 ml/minute/ 1.73m2 at two consecutive determinations (one GFR result from the screening visit labs and another GFR result from a prior laboratory determination and/or an unscheduled visit to confirm that the GFR is truly within the correct range.)

Exclusion Criteria:

* Prior use of experimental drug, MK-0677
* Subject has been diagnosed with neuromuscular or neurological disease causing muscle weakness.
* Body mass index greater than 35 kg/m2, or morbid obesity
* Uncontrolled hypothyroidism, defined as an elevated serum thyroid stimulating hormone (TSH) and a free serum thyroxine (T4) less than the lower limit of normal, when tested at screening (Patients requiring thyroid replacement during the study may continue.)
* Uncontrolled hyperthyroidism, defined as a TSH less than the lower limit of normal and an elevated free T4, when tested at screening
* Hemoglobin < 10 Gm/dl at screening
* Elevated serum transaminases (alanine transaminase (ALT) and aspartate transaminase (AST). (≥2.0 times the upper limit of normal at screening)
* Elevated alkaline phosphatase (Alk Phos). (≥3.0 times the upper limit of normal at screening)
* Diabetes with one or more of the following:

  1. Poorly controlled diabetes as defined by a HbA1C >7.0% at screening
  2. Pre-proliferative and Proliferative diabetic retinopathy [To participate in this study, diabetic patients will need to have had a dilated ophthalmology exam or retinal photography within 12 months of enrollment. Individuals who already have extensive background retinopathy will need to have a dilated ophthalmology exam within the 3 months of enrollment. Patients with pre-proliferative or proliferative retinopathy will be excluded.]
  3. Unwilling or unable to check blood glucose at home at least daily
* Currently receiving a systemic corticosteroid dose of ≥10 mg prednisone. (The previous use, or current use, of a topical or inhaled corticosteroid is allowed.)
* Currently taking or previously on an anabolic steroid or growth hormone at any dose, or for any duration, during the 12 months prior to study entry.
* Significant end-organ disease, other than kidney disease, which, in the opinion of the investigator may pose an added risk to the patient, confound the study results, or impair the patient's ability to complete the trial.
* Any of the following disorders within 6 months prior to baseline:

  1. Acute coronary syndrome (e.g., myocardial infarction or unstable angina)
  2. Coronary artery intervention (e.g., coronary bypass graft [CABG], percutaneous transluminal coronary angioplasty [PTCA])
  3. Stroke or transient ischemic neurological disorder (e.g. transient ischemic attack [TIA])
* New or worsening signs or symptoms of coronary heart disease within the 3 months prior to baseline
* NYHA (New York Heart Association) Class III or IV congestive heart failure (definitions shown in Appendix A)
* Uncontrolled hypertension when checked at screening visit: as evidenced by >160 systolic and/or 100 diastolic (measured in dominant arm, after at least 5 minutes, sitting)
* Cancer, or diagnosis of malignancy within the last 5 years, except for adequately treated basal cell or squamous cell skin cancer, or adequately treated in situ cervical cancer
* Active carpal tunnel syndrome
* Patient is, in the opinion of the investigator, mentally or legally incapacitated such that informed consent cannot be obtained or such that adherence to the study procedures and dosing regimens is questionable
* Patient is, at study entry, a regular user (including "recreational use") of illicit drugs or had a recent history (within the last 5 years) of drug or alcohol abuse. (a drug screen will not be done, this information will be obtained by history)
* Patient plans to relocate during the study, rendering follow-up per protocol, impractical
* Patient is participating in, or has participated in, another study with an investigational drug within 30 days prior to signing the informed consent form.
* If female, patient must not be pregnant or nursing. Patient must be postmenopausal, surgically sterilized, or willing to take adequate contraceptive precautions (i.e. use double barrier methods).
* HIV positive (medical history review and patient report)
* Patient is on potent CYP3A4 Inhibitor or Inducer Drugs within one week of starting study drug

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Lean body weight. | 12 months
  N/A - Study Withdrawn

SECONDARY OUTCOMES:
Cytokine levels | 12 months
  N/A - Study Withdrawn
Hormone levels | 12 months
  N/A - Study Withdrawn
Nutritional status | 12 months
  N/A - Study Withdrawn
Quality of life | 12 months
  N/A - Study Withdrawn
Physical function | 12 months
  N/A - Study Withdrawn

CONTACTS AND LOCATIONS:
Overall Officials: Warren K. Bolton, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States